CLINICAL TRIAL: NCT04685889
Title: Clinical Evaluation of the Effect of Resin Infiltration Treatment on Hypomineralised Enamel Surfaces
Brief Title: Resin Infiltration Treatment for MIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Associated professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018/35
Record Dates: First submitted 2020-12-13; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Molar Incisor Hypomineralization; Enamel Hypoplasia; Enamel Caries; Anterior Teeth
Keywords: molar incisor hypomineralisation; resin infiltration; discoloration; enamel; lesion
MeSH Terms: conditions — Molar Hypomineralization; Dental Enamel Hypoplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icon Group (Active Comparator): Icon® resin infiltration treatment was performed on 58 permanent central teeth with MIH and evaluated before; immediately after; and 1, 3, and 6 months after the procedure.
  Interventions: Procedure: Resin infiltration
- Control Group (No Intervention): No treatment was performed on healthy teeth. However, similar to the treated teeth, 58 healthy permanent central teeth of the same individuals were evaluated before; immediately after; and 1, 3, and 6 months after the procedure.

INTERVENTIONS:
Procedure: Resin infiltration — A sufficient amount of HCl was applied to the lesion using the icon etch syringe included in the set and was allowed to sit for 2 minutes. After washing with water for 30 seconds, the tooth was dried using an air spray. Once the enamel surface appeared chalky, Icon® dry application was initiated.
  Ethanol was applied to the lesion using the Icon® dry syringe included in the set, and after 30 seconds it was dried using an air spray. Sufficient amount of resin infiltrant was applied to the lesion using the Icon® infiltrant syringe. The resin infiltrant was applied to the lesion surface by massaging with the tip of the syringe in circular movements for 3 minutes such that it penetrates the surface thoroughly. The resin infiltrant was polymerized for 40 seconds with a light device.
  Arms: Icon Group

SUMMARY:
The investigators aimed to evaluate changes in mineralisation degree, colour, and size of the lesion after Icon® in permanent teeth with MIH in 6 months.

DETAILED DESCRIPTION:
A total of 116 permanent central teeth of 37 patients were included in the study. Icon® was applied to teeth with MIH, while the healthy teeth received no treatment (control).

Group I : Icon® resin infiltration treatment was performed on 58 permanent central teeth with MIH and evaluated before; immediately after; and 1, 3, and 6 months after the procedure.

Group II (Control Group): No treatment was performed on healthy teeth. However, similar to the treated teeth, 58 healthy permanent central teeth of the same individuals were evaluated before; immediately after; and 1, 3, and 6 months after the procedure.

Lesions were evaluated before, immediately after, and 1, 3, and 6 months after treatment. Mineralisation degree of MIH lesions was evaluated using DIAGNOdent Pen, changes in the lesion colour and lesion size were evaluated using VITA EasyShade and the cross polarization technique, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Molar incisor hypomineralisation on the labial surface of permanent central teeth Least one of the labial surface of the permanent anterior teeth were affected by MIH.

Exclusion Criteria:

* Dental caries and filling on anterior teeth.
* Dental anomaly on anterior teeth.
* Undergoing orthodontic treatment.
* Periodontal diseases.
* Cognitive and behavioural problems.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2018-06-23 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in the Mineralisation degree | Baseline (before resin infiltration), immediately after resin infiltration, 1 month later, 3 months later, 6 months later
  MIH lesions was evaluated using DIAGNOdent Pen (laser fluorescence)
Changes in the lesion colour | Baseline (before resin infiltration), immediately after resin infiltration, 1 month later, 3 months later, 6 months later
  Changes in the MIH lesions colour was evaluated using VITA EasyShade (Spectrophotometers are equipped with sensors that can measure in many wavelengths)
Lesion size evaluated using cross polarization technique | Baseline (before resin infiltration), immediately after resin infiltration, 1 month later, 3 months later, 6 months later
  Changes in the MIH lesions size was evaluated using cross polarization technique

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Altan, assoc. prof., Study Director — Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pediatric Dentistry; Rabia Erağca Yılmaz, Msc. Dt., Principal Investigator — Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576
- [Background] Jeremias F, de Souza JF, Silva CM, Cordeiro Rde C, Zuanon AC, Santos-Pinto L. Dental caries experience and Molar-Incisor Hypomineralization. Acta Odontol Scand. 2013 May-Jul;71(3-4):870-6. doi: 10.3109/00016357.2012.734412. Epub 2013 Jan 28. PMID 23351220
- [Background] Jalevik B, Noren JG. Enamel hypomineralization of permanent first molars: a morphological study and survey of possible aetiological factors. Int J Paediatr Dent. 2000 Dec;10(4):278-89. doi: 10.1046/j.1365-263x.2000.00210.x. PMID 11310241
- [Background] Fearne J, Anderson P, Davis GR. 3D X-ray microscopic study of the extent of variations in enamel density in first permanent molars with idiopathic enamel hypomineralisation. Br Dent J. 2004 May 22;196(10):634-8; discussion 625. doi: 10.1038/sj.bdj.4811282. PMID 15153976
- [Background] Dantas-Neta NB, Soares Figueiredo M, Lima CCB, Bendo CB, Matos de Andrade EM, Lima MDM, Pordeus IA, Paiva SM. Factors associated with molar-incisor hypomineralisation in schoolchildren aged 8-10 years: a case-control study. Int J Paediatr Dent. 2018 Nov;28(6):570-577. doi: 10.1111/ipd.12412. Epub 2018 Jul 17. PMID 30019508
- [Background] Cho SY, Ki Y, Chu V. Molar incisor hypomineralization in Hong Kong Chinese children. Int J Paediatr Dent. 2008 Sep;18(5):348-52. doi: 10.1111/j.1365-263X.2008.00927.x. Epub 2008 Jul 10. PMID 18637048
- [Background] Dietrich G, Sperling S, Hetzer G. Molar incisor hypomineralisation in a group of children and adolescents living in Dresden (Germany). Eur J Paediatr Dent. 2003 Sep;4(3):133-7. PMID 14529334
- [Background] Heitmuller D, Thiering E, Hoffmann U, Heinrich J, Manton D, Kuhnisch J, Neumann C, Bauer CP, Heinrich-Weltzien R, Hickel R; GINIplus Study Group. Is there a positive relationship between molar incisor hypomineralisations and the presence of dental caries? Int J Paediatr Dent. 2013 Mar;23(2):116-24. doi: 10.1111/j.1365-263X.2012.01233.x. Epub 2012 Mar 2. PMID 22384801
- [Background] Kuscu OO, Caglar E, Aslan S, Durmusoglu E, Karademir A, Sandalli N. The prevalence of molar incisor hypomineralization (MIH) in a group of children in a highly polluted urban region and a windfarm-green energy island. Int J Paediatr Dent. 2009 May;19(3):176-85. doi: 10.1111/j.1365-263X.2008.00945.x. Epub 2008 Nov 11. PMID 19016928
- [Background] Soviero V, Haubek D, Trindade C, Da Matta T, Poulsen S. Prevalence and distribution of demarcated opacities and their sequelae in permanent 1st molars and incisors in 7 to 13-year-old Brazilian children. Acta Odontol Scand. 2009;67(3):170-5. doi: 10.1080/00016350902758607. PMID 19253064
- [Background] Martos J, Gewehr A, Paim E. Aesthetic approach for anterior teeth with enamel hypoplasia. Contemp Clin Dent. 2012 Apr;3(Suppl 1):S82-5. doi: 10.4103/0976-237X.95112. PMID 22629075
- [Background] Muniz RSC, Carvalho CN, Aranha ACC, Dias FMCS, Ferreira MC. Efficacy of low-level laser therapy associated with fluoride therapy for the desensitisation of molar-incisor hypomineralisation: Randomised clinical trial. Int J Paediatr Dent. 2020 May;30(3):323-333. doi: 10.1111/ipd.12602. Epub 2019 Dec 23. PMID 31808584
- [Background] Meyer-Lueckel H, Paris S, Kielbassa AM. Surface layer erosion of natural caries lesions with phosphoric and hydrochloric acid gels in preparation for resin infiltration. Caries Res. 2007;41(3):223-30. doi: 10.1159/000099323. PMID 17426404
- [Background] William V, Messer LB, Burrow MF. Molar incisor hypomineralization: review and recommendations for clinical management. Pediatr Dent. 2006 May-Jun;28(3):224-32. PMID 16805354
- [Background] Paris S, Meyer-Lueckel H, Kielbassa AM. Resin infiltration of natural caries lesions. J Dent Res. 2007 Jul;86(7):662-6. doi: 10.1177/154405910708600715. PMID 17586715
- [Background] Zandona AF, Zero DT. Diagnostic tools for early caries detection. J Am Dent Assoc. 2006 Dec;137(12):1675-84; quiz 1730. doi: 10.14219/jada.archive.2006.0113. PMID 17138712
- [Background] Lussi A, Hibst R, Paulus R. DIAGNOdent: an optical method for caries detection. J Dent Res. 2004;83 Spec No C:C80-3. doi: 10.1177/154405910408301s16. PMID 15286128
- [Background] Robertson AJ, Toumba KJ. Cross-polarized photography in the study of enamel defects in dental paediatrics. J Audiov Media Med. 1999 Jun;22(2):63-70. doi: 10.1080/014051199102179. PMID 10628000
- [Background] Knosel M, Eckstein A, Helms HJ. Durability of esthetic improvement following Icon resin infiltration of multibracket-induced white spot lesions compared with no therapy over 6 months: a single-center, split-mouth, randomized clinical trial. Am J Orthod Dentofacial Orthop. 2013 Jul;144(1):86-96. doi: 10.1016/j.ajodo.2013.02.029. PMID 23810050
- [Background] Farah RA, Drummond BK, Swain MV, Williams S. Relationship between laser fluorescence and enamel hypomineralisation. J Dent. 2008 Nov;36(11):915-21. doi: 10.1016/j.jdent.2008.07.012. Epub 2008 Sep 10. PMID 18786755
- [Background] Johnston WM, Reisbick MH. Color and translucency changes during and after curing of esthetic restorative materials. Dent Mater. 1997 Mar;13(2):89-97. doi: 10.1016/s0109-5641(97)80017-6. PMID 9467310
- [Background] Rocha Gomes Torres C, Borges AB, Torres LM, Gomes IS, de Oliveira RS. Effect of caries infiltration technique and fluoride therapy on the colour masking of white spot lesions. J Dent. 2011 Mar;39(3):202-7. doi: 10.1016/j.jdent.2010.12.004. Epub 2010 Dec 21. PMID 21172402
- [Background] Yetkiner E, Wegehaupt F, Wiegand A, Attin R, Attin T. Colour improvement and stability of white spot lesions following infiltration, micro-abrasion, or fluoride treatments in vitro. Eur J Orthod. 2014 Oct;36(5):595-602. doi: 10.1093/ejo/cjt095. Epub 2014 Jan 2. PMID 24385411
- [Background] Shivanna V, Shivakumar B. Novel treatment of white spot lesions: A report of two cases. J Conserv Dent. 2011 Oct;14(4):423-6. doi: 10.4103/0972-0707.87217. PMID 22144817
- [Background] Ruyter IE, Nilner K, Moller B. Color stability of dental composite resin materials for crown and bridge veneers. Dent Mater. 1987 Oct;3(5):246-51. doi: 10.1016/S0109-5641(87)80081-7. No abstract available. PMID 3479360
- [Background] Johnston WM, Kao EC. Assessment of appearance match by visual observation and clinical colorimetry. J Dent Res. 1989 May;68(5):819-22. doi: 10.1177/00220345890680051301. PMID 2715476
- [Background] Khanna R, Chandra A, Singh RK. Quantitative evaluation of masking effect of resin infiltration on developmental defects of enamel. Quintessence Int. 2020;51(6):448-455. doi: 10.3290/j.qi.a44493. PMID 32368763
- [Derived] Altan H, Yilmaz RE. Clinical evaluation of resin infiltration treatment masking effect on hypomineralised enamel surfaces. BMC Oral Health. 2023 Jul 3;23(1):444. doi: 10.1186/s12903-023-03140-6. PMID 37400849